CLINICAL TRIAL: NCT02097251
Title: An Open-Label Treatment Protocol With UX003 Recombinant Human Beta-glucuronidase (rhGUS) Enzyme Replacement Therapy for an Advanced Stage Mucopolysaccharidosis Type 7 (MPS 7) Patient
Brief Title: An Open-Label Treatment Protocol With UX003 rhGUS Enzyme Replacement Therapy for an Advanced Stage MPS 7 Patient
Status: No longer available | Type: Expanded Access
Sponsor: Joyce Fox (Other)
Collaborators: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor-Investigator, Joyce Fox, Chief of Medical Genetics at Cohen Children's Medical Center, Northwell Health
Organization: Northwell Health (Other)
Other Study IDs: 13-606A
Record Dates: First submitted 2014-03-24; First posted 2014-03-27 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-02

CONDITIONS: Mucopolysaccharidosis Type 7
Keywords: Mucopolysaccharidosis Type 7; Sly syndrome; UX003; Enzyme Replacement Therapy; rare disease; Lysosomal Storage Disease; metabolic disorder
MeSH Terms: conditions — Mucopolysaccharidosis VII; Rare Diseases; Lysosomal Storage Diseases; Metabolic Diseases | interventions — vestronidase alfa

INTERVENTIONS:
Drug: UX003 — Open Label
  Other Names: recombinant human beta glucuronidase; rhGUS

SUMMARY:
Emergency access granted to treat a single patient with advanced Mucopolysaccharidosis Type 7 with UX003 Recombinant Human Beta-glucuronidase (rhGUS) Enzyme Replacement Therapy via IV administration every other week (QOW) for up to 144 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 1 specific patient
* Confirmed diagnosis of MPS 7 based on leukocyte or fibroblast glucuronidase enzyme assay or genetic testing confirming diagnosis.
* Written informed consent of parent(s) or legal guardian(s)

Sex: Male
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Cohen Children's Medical Center, New Hyde Park, New York, United States